CLINICAL TRIAL: NCT06728033
Title: Comparison of Perioperative Analgesic Effects of Preoperative Supra-inguinal Fascia Iliaca Compartment Block and Intravenous Tramadol in Hip Fracture: A Randomized Controlled Trial
Brief Title: Fascia Iliaca Compartment Block and Tramadol for Analgesia in Hip Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCH20241201
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hip Fractures; Ultrasound-guided Nerve Block; Perioperative Analgesia
Keywords: Hip Fractures; Supra-inguinal Fascia Iliaca compartment Block; Tramadol
MeSH Terms: conditions — Hip Fractures | interventions — Tramadol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As the clinical management differs between groups, researchers, participants, and clinical staff will be aware of the group allocations; however, follow-up personnel, outcome assessors, and statisticians will remain blinded to group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SiFICB Group (Experimental): Participants will receive an ultrasound-guided SiFICB above the inguinal ligament with 40 ml of 0.25% ropivacaine.
  Interventions: Other: supra-inguinal fascia iliaca compartment block
- Tramadol Group (Active Comparator): Participants will receive intravenous tramadol at a dose of 2 mg/kg
  Interventions: Drug: Tramadol

INTERVENTIONS:
Other: supra-inguinal fascia iliaca compartment block — Supra-inguinal fascia iliaca compartment block with 40 ml of 0.25% ropivacaine
  Arms: SiFICB Group
Drug: Tramadol — intravenous tramadol at a dose of 2 mg/kg
  Arms: Tramadol Group

SUMMARY:
Hip fractures are a growing public health concern globally due to the aging population, with high incidence and significant mortality rates one year post-fracture. Effective pain management is critical to improving outcomes and accelerating recovery. Tramadol, a widely used intravenous analgesic, has dual opioid and non-opioid mechanisms but is associated with side effects, such as nausea, dizziness, and respiratory depression, necessitating careful monitoring in hip fracture patients.

The supra-inguinal fascia iliaca compartment block (SiFICB) offers a promising alternative, targeting key nerves to achieve effective analgesia through ultrasound-guided delivery of local anesthetics. SiFICB minimizes side effects and improves pain control by accurately blocking the femoral, lateral femoral cutaneous, and obturator nerves. While its postoperative benefits are well-documented, its efficacy in managing preoperative pain from hip fractures remains underexplored.

This study hypothesizes that ultrasound-guided SiFICB provides superior perioperative analgesia compared to intravenous tramadol. A prospective randomized controlled trial will evaluate the analgesic efficacy of SiFICB, using the numerical rating scale (NRS) to assess pain, aiming to improve the management of hip fracture-related pain and patient outcomes.

DETAILED DESCRIPTION:
Background With the global aging population, the incidence of hip fractures continues to rise. In the United States, over 300,000 cases occur annually among individuals aged 65 years or older. The incidence of hip fractures in Europe ranges between 307 and 1269 per 100,000 population. Mortality rates one year after a hip fracture are alarmingly high, ranging from 19.7% to 34.8%, making hip fractures a significant public health issue. It is estimated that the global number of hip fracture cases will increase to 2.6-7.3 million by 2025 and 4.5-21.3 million by 2050 . Optimizing treatment pathways for hip fractures, promoting accelerated postoperative recovery, and improving patient outcomes are therefore critical.

Early pain management intervention can alleviate pain, reduce anxiety, improve sleep, and significantly decrease complications and mortality associated with hip fractures . Currently, intravenous tramadol is a commonly used analgesic. Tramadol, a synthetic opioid, acts as a μ-opioid receptor agonist with weak affinity and inhibits serotonin (5-HT) and norepinephrine (NE) reuptake, exerting dual analgesic effects . It is increasingly replacing high-affinity opioids for the treatment of moderate-to-severe acute and chronic pain globally. However, tramadol has adverse effects, including sweating, dizziness, nausea, vomiting, appetite loss, urinary retention, and risks of addiction, misuse, and respiratory depression. Its use in hip fracture patients requires close monitoring to manage adverse effects promptly.

The pain associated with hip fractures arises from noxious stimulation of free nerve endings transmitting nociceptive and proprioceptive signals. The nerves innervating the hip skin originate from the lumbar plexus, including the femoral nerve and lateral femoral cutaneous nerve. The anterior hip joint capsule receives sensory input from the femoral and obturator nerves. Pain receptors in the anterior capsule are most densely distributed in the superior portion, while they are sparse in the posterior capsule and ligaments surrounding the hip joint.

Based on this anatomical understanding, a Supra-inguinal fascia iliaca compartment block (SiFICB) above the inguinal ligament can effectively block the femoral and lateral femoral cutaneous nerves. The spread of local anesthetics medially in the fascia iliaca compartment can also block the obturator nerve, achieving analgesia. However, fascia iliaca blocks can have adverse effects, including inadequate localization leading to poor efficacy, quadriceps weakness due to femoral nerve blockade, and local anesthetic toxicity. Ultrasound guidance can ensure accurate delivery of local anesthetics into the fascia iliaca compartment, allowing for lower concentrations and reduced adverse effects. Although studies have reported the efficacy of ultrasound-guided fascia iliaca blocks for postoperative pain relief after hip surgeries , their impact on preoperative pain caused by fracture displacement or friction of fracture ends remains underexplored.

The investigators hypothesize that an ultrasound-guided SiFICB above the inguinal ligament provides superior perioperative analgesia compared with intravenous tramadol, the current standard of care in orthopedic trauma. To test this hypothesis, the investigators design a prospective randomized controlled trial in patients undergoing hip fracture surgery, using the numerical rating scale (NRS) as the primary outcome to assess pain, to evaluate the perioperative analgesic efficacy of ultrasound-guided SiFICB by comparison to intravenous tramadol in patients with hip fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of hip fracture
* Aged >18 years, of any gender
* Provide signed and dated written informed consent before formal enrollment in the study.

Exclusion Criteria:

* Allergic to tramadol or ropivacaine
* Unable to cooperate with the study for any reason, such as language comprehension issues, psychiatric disorders, severe hearing impairments, or communication barriers
* Unsuitable for the trial by the investigator based on clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting numerical rating scale (NRS) pain scores preoperatively | 7 days postperatively
  The Numerical Rating Scale (NRS) is a tool for assessing pain intensity, allowing patients to rate their pain on a scale from 0 to 10, where 0 represents "no pain," 10 represents "the worst pain imaginable," and pain levels are categorized as 0 (no pain), 1-3 (mild pain), 4-6 (moderate pain), and 7-10 (severe pain).

SECONDARY OUTCOMES:
Incidence of severe complications | 7 days postperatively
  Mortality and the overall incidence of severe complications are classified into five grades: Grade I (fully resolved with temporary treatment, e.g., postoperative nausea and vomiting), Grade II (prolonged hospital stay required, e.g., pneumonia requiring antibiotic treatment), Grade III (life-threatening events requiring intervention with recovery during hospitalization, e.g., deep vein thrombosis), Grade IV (significant long-term harm, e.g., postoperative cognitive dysfunction), and Grade V (death within 30 days postoperatively).
Resting NRS pain scores postoperatively | 3 days after surgery
  Resting NRS pain scores on postoperative days 1, 2, and 3
Movement NRS pain scores postoperatively | 3 days after surgery
  Movement NRS pain scores on postoperative days 1, 2, and 3
Total perioperative morphine consumption | 7 days postperatively
  Morphine is used as a rescue measure for acute pain. When a patient's resting NRS pain score exceeds 4, 5 mg of morphine can be administered intravenously. If the effect is insufficient, an additional 5 mg may be given after 30 minutes, with a maximum daily dose of 20 mg.
Time to initiation of functional exercise | 30 days postperatively
  Duration from admission to the first mobilization, pre- or postoperatively (days)
Total length of hospital stay | 30 days postperatively
  Duration from admission to discharge (days)
Postoperative hospital stay | 30 days postperatively
  Duration from surgery to discharge (days)
Total hospitalization costs | 7 days after discharge
  Total hospitalization costs

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after de-identification.The shared data will include de-identified individual participant data, and metadata supporting the primary and secondary outcomes, as well as the study protocol.Data will be available beginning 6 months after publication of the main study results and ending 3 years following publication.
  Requests for data sharing should be directed to the corresponding author (liaoren7733@163.com). Upon approval of a formal proposal, a data-sharing agreement will be signed, and access will be granted through a secure data-sharing platform.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 months after publication of the main study results and ending 3 years following publication.
Access Criteria: Requests for data sharing should be directed to the corresponding author (liaoren7733@163.com).